CLINICAL TRIAL: NCT02054221
Title: Compare Results of Mitral Valve Replacement or Repair in the Surgical Treatment of Obstructive Hypertrophic Cardiomyopathy With Severe Mitral Insufficiency.
Brief Title: Surgical Treatment of Hypertrophic Obstructive Cardiomyopathy With Severe Mitral Insufficiency.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HOCM - 95; 1957 (Other: NRICP)
Record Dates: First submitted 2013-12-27; First posted 2014-02-04 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: hypertrophic cardiomyopathy; mitral valve
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- extended myectomy + MVreplacement (Other): Procedure: extended myoectomy, mitral valve surgery
  Will be included in a group of 41 patients with obstructive hypertrophic cardiomyopathy and severe mitral insufficiency. Intraoperatively for all patients will be executed TEE to calculate the volume of excision. All patients will be performed extended myoectomy with full isscheniem subvalvular apparatus and mitral valve replacement.
  Evaluation results will be made myoectomy as TEE and direct tensiometer.
  Interventions: Procedure: myoectomy; Procedure: Mitral valve surgery
- extended myectomy + MVrepair (Other): Procedure: extended myoectomy, mitral valve surgery
  Will be included in a group of 41 patients with obstructive hypertrophic cardiomyopathy and severe mitral insufficiency. Intraoperatively for all patients will be executed TEE to calculate the volume of excision. All patients will be performed extended myoectomy which supplemented resection and release of the papillary muscles and the mitral valve repair. Results of mitral valve repair will be more appreciated intraoperatively. In case of unsatisfactory MV repair will reconnect the device artificial circulation and mitral valve replacement. There after, patients will be moved to the first group.
  Evaluation results will be made myoectomy as TEE and direct tensiometer .
  Interventions: Procedure: myoectomy; Procedure: Mitral valve surgery

INTERVENTIONS:
Procedure: myoectomy — The scheme of Extended septal myectomy: Two parallel incisions were made into the septal bulge and connected to remove the muscle mass. Myectomy was extended to the base of the papillary muscles, when midseptal thickening was present. The papillary muscles were grasped and pushed medially to visualize the abnormal connections between the papillary muscles and the anterior wall of the ventricle. A blade was used to divide the thickened abnormal attachments. A pituitary rongeur may be used to resect a portion of the junction of the papillary and lateral wall. This reduces the diameter of the papillary muscle and allows for posterior displacement of the anterior mitral leaflet. Division of abnormal attachments and thinning of the papillary muscles is critical for the treatment of SAM.
  Other Names: Extended myoectomy
Procedure: Mitral valve surgery — 41 patients will be performed mitral valve replacement with complete excision of the subvalvular apparatus.
  Other Names: mitral valve replacement
  Arms: extended myectomy + MVreplacement
Procedure: Mitral valve surgery — 41 patients will be performed mitral valve repair. Results of mitral valve repair will be more appreciated intraoperatively. In case of unsatisfactory MV repair will reconnect the device artificial circulation and mitral valve replacement. There after, patients will be moved to the first group.
  Other Names: mitral valve repair
  Arms: extended myectomy + MVrepair

SUMMARY:
Compare the results of reconstruction and mitral valve replacement in the surgical treatment of obstructive hypertrophic cardiomyopathy with severe mitral insufficiency.

DETAILED DESCRIPTION:
Many years myoectomy for Morrow was the gold standard in the treatment of obstructive hypertrophic cardiomyopathy. Currently more retrospective data in the literature about the good results the extended septal myectomy. But the question remains what is best for patients with obstructive hypertrophic cardiomyopathy and severe mitral insufficiency: use extended myoectomy with mitral valve repair a or replacement.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign Informed Consent and Release of Medical Information forms
* Age ≥ 18 years
* obstructive hypertrophic cardiomyopathy
* surgically significant mitral insufficiency
* II-IV (NYHA),
* average systolic pressure gradient greater than 50 mm Hg. Art. at rest;
* basal or medium ventricular obstruction

Exclusion Criteria:

* Related defect of the aortic valve;
* Organic mitral valve disease (dysplasia, rheumatic fever, infective endocarditis);
* Surgically significant coronary artery lesions;
* Patients requiring implantation of a cardioverter-defibrillator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The function of the mitral valve (mitral regurgitation return, prosthesis dysfunction) | one year

SECONDARY OUTCOMES:
The pressure gradient in the output section of the left ventricle | one year

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr V Bogachev-Prokophiev, PhD, Principal Investigator — Meshalkin Research Institute of Pathology of Circulation
Locations (1):
- Novosibirsk State Research Institute of Circulation Pathology, Novosibirsk, Novosibirsk Territory, Russia

REFERENCES:
- [Background] Surgical Treatment of Hypertrophic Obstructive Cardiomyopathy With severe Mitral regurgitation
- [Derived] Bogachev-Prokophiev A, Afanasyev A, Zheleznev S, Fomenko M, Sharifulin R, Kretov E, Karaskov A. Mitral valve repair or replacement in hypertrophic obstructive cardiomyopathy: a prospective randomized study. Interact Cardiovasc Thorac Surg. 2017 Sep 1;25(3):356-362. doi: 10.1093/icvts/ivx152. PMID 28575282